CLINICAL TRIAL: NCT05016921
Title: Transcutaneous Magnetic Stimulation of the Stellate Ganglion to Treat Ventricular Tachycardia
Brief Title: TcMS to Treat Ventricular Tachycardia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Alternate study pursued
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 849193
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcutaneous magnetic stimulation (Experimental): Transcutaneous magnetic stimulation targeting the stellate ganglion
  Interventions: Device: TcMS

INTERVENTIONS:
Device: TcMS — Transcutaneous magnetic stimulation targeting the stellate ganglion

SUMMARY:
Open label study of transcutaneous magnetic stimulation targeting the stellate ganglion in patients with ventricular tachycardia

ELIGIBILITY:
Inclusion Criteria:

* Age >18years
* Documented ventricular tachycardia within the preceding 72 hours

Exclusion Criteria:

* Pregnancy
* Implanted ventricular assist device
* Metal implanted in heard or neck (except the mouth)
* Implanted medication pumps
* Cochlear implant
* Implanted brain stimulator
* Ocular implant
* History of malignancy in the region of stimulation (neck)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Ventricular Tachycardia | 0-72 hours after enrollment
  Burden (number of episodes) of ventricular tachycardia

SECONDARY OUTCOMES:
Non sustained ventricular tachycardia | 0-72 hours after enrollment
  Burden (number of episodes) of ventricular tachycardia
Discomfort | Assessed immediately following stimulation
  Discomfort experienced during stimulation (on scale of 0-10) reported by patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No